CLINICAL TRIAL: NCT06381037
Title: Quality of Life and Psychological Strengths of Older People: Assessment and Intervention
Brief Title: Quality of Life and Psychological Strengths of Older People
Acronym: QUALIFRAG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PID2021-127986OB-I00
Record Dates: First submitted 2023-12-11; First posted 2024-04-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Quality of Life; Skills, Coping
Keywords: Elderly; Quality of life; Strengths
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Intervention Model Description: Quantitative, observational and longitudinal study with three measurements (pre-intervention, post-intervention and monitoring).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group is given the workshop "How to improve your strengths and quality of life".
  Interventions: Behavioral: "How to improve your strengths and quality of life".
- Control group (No Intervention): The control group is not given the workshop "How to improve your strengths and quality of life".

INTERVENTIONS:
Behavioral: "How to improve your strengths and quality of life". — The intervention program "How to improve your strengths and quality of life" consists of 9 individual sessions. The sessions take place weekly, so the total duration of the program is 9 weeks. Each session lasts approximately 1 hour. The sessions will be held both in person and online.
  The sessions are as follows:
  * Session 0. Presentation of the programme
  * Session 1. Introduction to quality of life and personal strengths
  * Session 2. Self-realisation
  * Session 3. Pleasure and gratitude
  * Session 4. Autonomy and control
  * Session 5. Family functioning and assertive communication
  * Session 6. Resilience
  * Session 7. Experiential acceptance
  * Session 8. Closing and farewell
  Arms: Experimental group

SUMMARY:
Older adults have psychological strengths that promote psychological well-being and reduce distress (depression or anxiety) and loneliness, enhancing their quality of life (QoL). These strengths can play a key role in a psychological intervention programme to promote QoL.

Ageing and stress may increase the likelihood of illness in older people. When social policies and values, such as ageism and age-based discrimination, are added to this, older people are perceived as one of the most vulnerable groups in the population. The novelty of the study focuses on the paradigm shift regarding ageing, from the traditional model of decline associated with older people, in which ageing is associated with illness, functional decline and dependence, to a more positive view focused on personal strengths to cope with adversity, and how this relates to psychological well-being, emotional distress and QoL. The first and main reason for conducting this research is the scarcity of studies based on the model of strengths or gains in relation to ageing.

Therefore, the relevance of this study lies, on the one hand, in offering a change of perspective on old age, from a negative view (illness or vulnerability) to an approach based on strengths, and on the other hand, in gaining a deeper understanding of the strengths of older people, the associated factors and the role they play in cushioning adversity, such as in the COVID-19 pandemic. Most older people remain healthy, independent and enjoy high levels of well-being and QoL, with factors such as resilience cushioning the consequences of stress and ageing.

In this vein, it has been shown that age strengthens the ability to distance oneself from stressful situations and re-evaluate them positively, and older people report greater emotional well-being compared to younger adults. Furthermore, it is well known that having good social support seems to have long-term health benefits. Some recent studies related to the pandemic show that older people, despite being the most threatened by the situation, had lower levels of anxiety and depression compared to younger people, contrary to expectations. Furthermore, coping strategies, such as resilience and social support, are mediating factors in the well-being of older people exposed to COVID-19.

Psychology, and psychogerontology in particular, is responsible for designing interventions aimed at increasing the likelihood of successful ageing. In fact, managing emotions is essential for people's health, well-being and QoL. In this sense, the emergence of positive psychology represents a change in therapeutic and rehabilitation processes. This psychological trend leaves behind a model based mainly on negative aspects and loss, in order to enhance human qualities that can act as buffers against adversity. In this way, a shift in focus is established, suggesting that in addition to trying to alleviate pathological aspects, it is equally important to find people's qualities or virtues in order to achieve greater QoL.

COVID-19 has led to older people being portrayed as a homogeneous group, even though increased life expectancy means that this is the longest stage of life, with studies reflecting the great diversity of older people. They are repeatedly portrayed as vulnerable, with messages that convey paternalism ('our elders') and overprotection, despite scientific literature indicating that this can have serious consequences. Throughout their lives, older people have had to face adversity, which they have been able to overcome or accept thanks to psychological strengths such as resilience, acceptance and gratitude, among others.

DETAILED DESCRIPTION:
The intervention program "How to improve your strengths and quality of life" consists of 9 individual sessions. The sessions take place weekly, so the total duration of the program is 9 weeks. Each session lasts approximately 1 hour. The sessions will be held both in person and online.

Following the principles of the psychoeducational therapy and Positive Psychology, this program is focused on the enhancement of personal strengths and quality of life of the elderly. Specifically, during the sessions, the following topics will be worked on: resilience, gratitude, acceptance, family functioning and quality of life in its different dimensions (control, autonomy, pleasure and self-fulfillment).

The sessions are as follows:

* Session 0. Presentation of the programme.
* Session 1. Introduction to quality of life and personal strengths.
* Session 2. Self-realisation.
* Session 3. Pleasure and gratitude.
* Session 4. Autonomy and control.
* Session 5. Family functioning and assertive communication.
* Session 6. Resilience.
* Session 7. Experiential acceptance.
* Session 8. Closing and farewell.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 60 years of age.
* Residing in Spain.
* Not having a diagnosed neurological disease or severe psychopathological disorder, or other ailment that is incompatible with the understanding of the questionnaires or the intervention program.
* Acceptance and signature of the informed consent.

Exclusion Criteria:

* Do not comply with the established age range.
* Present an ailment that makes them unable to respond to the questionnaire.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life | Through study completion, and average of 4 years.
  Quality of life will be evaluated with Quality of Life Questionnaire for the Elderly (CASP-12)
  Scale values: 1 (sometimes), 2, 3, 4 (never).
  Interpretation: the higher the score, the greater the quality of life of the person being assessed.
Psychological wellbeing | Through study completion, and average of 4 years.
  Psychological wellbeing will be evaluated with Ryff's Psychological Wellbeing Scale.
  Scale values: 1 (very inadequate to describe me), 2 (quite inadequate to describe me), 3 (some inadequate to describe me), 4 (some adequate to describe me), 5 (quite adequate to describe me), 6 (very adequate to describe me).
  Interpretation: the higher the score, the greater the psychological wellbeing of the person being assessed.
Loneliness | Through study completion, and average of 4 years.
  Loneliness will be evaluated with Three-Item Loneliness Scale.
  Scale values: 1 (hardly ever, 2 (some of the time), 3 (often).
  Interpretation: the higher the score, the greater the loneliness of the person being assessed.
Anxiety and depression Anxiety and depression | Through study completion, and average of 4 years.
  Anxiety and depression will be evaluated with Hospital Anxiety and Depression Scale.
  Scale values: values 2-4. The meaning of the values are different for each item.
  Interpretation: the higher the score, the greater the anxiety and depression of the person being assessed.
Gratitude | Through study completion, and average of 4 years.
  Gratitude will be evaluated with the short form of the Values in Action Inventory of Strengths (VIA-IS).
  Scale values: 1 (very different from me), 2 (somewhat different from me), 3 (neutral), 4 (somewhat similar to me), 5 (very similar to me).
  Interpretation: the higher the score, the greater the gratitude of the person being assessed.
Experiential acceptance | Through study completion, and average of 4 years.
  Experiential acceptance will be evaluated with the Acceptance and Action Questionnaire II.
  Scale values: 1 (never true), 2 (very seldom true), 3 (seldom true), 4 (sometimes true), 5 (frequently true), 6 (almost always true), 7 (always true).
  Interpretation: the higher the score, the greater the experiential acceptance of the person being assessed.
Resilience | Through study completion, and average of 4 years.
  Resilience will be evaluated with the Brief Resilient Coping Scale (BRCS).
  Scale values: 1 (it does not reflect a typical reaction in my), 2, 3, 4, 5 (it does reflect a typical reaction in my).
  Interpretation: the higher the score, the greater the resilience of the person being assessed.
Family functioning | Through study completion, and average of 4 years.
  Family functioning will be evaluated with the APGAR familiar.
  Scale values:0 (never), 1 (rarely), 2 (sometimes), 3 (almost always), 4 (always).
  Interpretation: the higher the score, the greater the family functioning of the person being assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- San Pablo CEU University (Campus Montepríncipe), Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available from August 2026.

DOCUMENTS (2):
  • Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT06381037/SAP_000.pdf
  • Informed Consent Form (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT06381037/ICF_001.pdf